CLINICAL TRIAL: NCT05658458
Title: A Phase IV Interventional Post Approval Trial to Investigate Effectiveness and Safety of Vericiguat Therapy in Indian Patients With Chronic Heart Failure With Reduced Ejection Fraction After a Worsening Heart Failure Event.
Brief Title: A Study to Learn How Well the Drug Vericiguat Works and How Safe it is Under Real World Conditions in Indian Participants After Worsening of a Long-term Heart Condition in Which the Left Side of the Heart Does Not Pump Blood as Well as it Should (Chronic Heart Failure With Reduced Ejection Fraction)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22144
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Chronic Heart Failure With Reduced Ejection Fraction; Worsening Heart Failure
MeSH Terms: interventions — vericiguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vericiguat therapy (Experimental): Adult participants with chronic HFrEF who are naïve to vericiguat and will be prescribed vericiguat as per local label by their treating physician (cardiologists).
  Interventions: Drug: Vericiguat (Verquvo, BAY1021189)

INTERVENTIONS:
Drug: Vericiguat (Verquvo, BAY1021189) — The recommended starting dose of vericiguat is 2.5 mg once daily, taken with food. The dose of vericiguat would be doubled approximately every 2 weeks to reach the target maintenance dose of 10 mg once daily, as tolerated by the participant.

SUMMARY:
Researchers are looking for a better way to treat people who have chronic heart failure with reduced ejection fraction (HFrEF).

HFrEF is a long-term condition where the left side of the heart does not pump blood out to the body as well as it should. Blood and fluid may collect in the lungs, blood vessels, and tissues causing shortness of breath or tiredness. Over time, heart failure can lead to other serious medical conditions that may result in hospital stays and death. Despite various available treatments for long-term HFrEF, people may experience worsening of their condition, called worsening heart failure events. Worsening heart failure events require the patient to either stay in the hospital or receive special treatment to remove excess water from the body.

The drug vericiguat works by increasing the activity of an enzyme called soluble guanylate cyclase (sGC). The sGC enzyme helps to regulate the heart and blood circulation. Vericiguat was recently approved in India for doctors to prescribe to people with HFrEF after they had a worsening heart failure event, with a request to specifically gather information on vericiguat therapy in Indians.

Therefore, the main purpose of this study is to learn more about how well vericiguat works in Indian people with HFrEF who receive vericiguat after a worsening heart failure event. Work well means to prevent:

* death due to heart and circulatory events, or
* hospital stays. Researchers will collect the number of participants treated with vericiguat who have either of this.

To find out how safe vericiguat is, researchers will also collect the number of participants who have medical problems during the study. Doctors keep track of all medical problems, even if they do not think the adverse events might be related to the study treatments.

The participants will take vericiguat as tablet by mouth and as prescribed by their doctors according to the local label.

Each participant will be in the study for approximately 1 year including a screening period of up to 1 month. Up to 8 visits to the study site are planned.

During the study, the study team will:

* check vital signs
* do physical examinations
* examine heart health using electrocardiogram ECG and if needed echocardiography
* take blood and urine samples

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged ≥18 years at the time point of signing ICF
* Has a history of chronic HF (NYHA class II-IV) on standard therapy before qualifying HF decompensation
* Has chronic HF with reduced LVEF (<45%) after a WHF event (defined as HF hospitalization or use of iv diuretics for HF [without hospitalization])
* Is capable of giving signed ICF and willing to comply with the study-related procedures
* Female participants in the following categories:

  * A female who is not of reproductive potential, defined as a female who either: (a) is postmenopausal (defined as at least 12 months with no menses in women ≥45 years of age); (b) has had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation/occlusion at least 6 weeks prior to Screening; or (c) has a congenital or acquired condition that prevents childbearing
  * A female who is of reproductive potential and agrees to avoid becoming pregnant while receiving the study drug and for 14 days after the last dose of the study drug by complying with one of the following: (a) practice abstinence from heterosexual activity or (b) use (and have her partner use) acceptable, highly effective contraception methods during heterosexual activity.

Exclusion Criteria:

* Is clinically unstable at the time of screening defined by:

  * Administration of any iv treatment within 24 hours until start of study intervention, and/or
  * SBP < 100 mmHg or symptomatic hypotension.
* Has concurrent or anticipated use of PDE5 inhibitors, or a sGC stimulator such as riociguat.
* Has known allergy or hypersensitivity to any sGC stimulator.
* Has severe hepatic insufficiency such as with hepatic encephalopathy.
* Has severe renal impairment with eGFR < 15 mL/min/1.73m*2 (calculated based on the MDRD equation) or on dialysis.
* Is pregnant or breast feeding or plans to become pregnant or to breastfeed during the course of the trial.
* Participated in another interventional clinical study and treatment with another investigational product ≤ 30 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Occurrence of the composite of CV death or first hospitalization due to HF | 14 days after end of treatment (EoT) visit (month 12) +1 week

SECONDARY OUTCOMES:
Occurrence of CV death | 14 days after end of treatment (EoT) visit (month 12) +1 week
Occurrence of first HF hospitalization | 14 days after end of treatment (EoT) visit (month 12) +1 week
Occurrence of the composite of death due to all causes or first HF hospitalization | 14 days after end of treatment (EoT) visit (month 12) +1 week
Occurrence of death due to all causes | 14 days after end of treatment (EoT) visit (month 12) +1 week
Occurrence of adverse events (AEs), serious adverse events (SAEs), study interventionrelated AEs will be listed | 14 days after end of treatment (EoT) visit (month 12) +1 week

CONTACTS AND LOCATIONS:
Locations (12):
- India (12):
  - Krishna Institute Of Medical Science, Secunderabad, Andhra Pradesh
  - Sanjivani Super Speciality Hospital, Ahmedabad, Gujarat
  - Rhythm Heart Institute, Vadodara, Gujarat
  - Lisie Hospital, Kochi, Kerala
  - Kokilaben Dhirubhai Ambani Hospital & Medical Research Insti, Mumbai, Maharashtra
  - Vijan Cardiac & Critical Care Centre, Nashik, Maharashtra
  - Max Super Speciality Hospital, Saket, New Delhi, National Capital Territory of Delhi
  - Safdarjung Hospital, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences, Bhubaneswar, Odisha
  - Deep Hospital, Ludhiana, Punjab
  - Apollo Hospital Tondiarpet, Chennai, Tamil N?du
  - Apollo Gleneagles Hospital Limited, Kolkata

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.